CLINICAL TRIAL: NCT02294045
Title: Analysis of Joint Sounds in the Diagnosis of Knee Disorders
Acronym: Joint
Status: Withdrawn | Type: Observational
Why Stopped: Unable to get the correct software.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Other Study IDs: 5120242
Record Dates: First submitted 2014-09-08; First posted 2014-11-19 (Estimated); Last update posted 2021-06-04 (Actual); Status verified 2021-06

CONDITIONS: Arthritis of Knee; Normal Knee; Knee Arthroscopy
Keywords: Knee; Healthy; arthroscopy; MRI; amplification; sounds; pre-operative; analyzing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical-noninvasive recording of sounds from the knees through a brief loaded range of motion. Description in phase 1 analytic but descriptive as well in phase 2. No samples other than a sound recording. The device is known microphone attached to the skin of the knee with elastic material. Sound recorded and analyzed on a lap top computer with Adobe software.

DETAILED DESCRIPTION:
There is a need for a less expensive and more universally available screening device for the knee, and other joint pathology. The equipment used for ultrasound is much less expensive and cumbersome than that of an x-ray or magnetic resonance imaging. The equipment we will use for the analysis of sound produced by the body itself is an order of magnitude less expensive than ultrasound; such as a laptop computer with currently available software and an inexpensive transducer. Analysis of sound has proved useful in Pulmonology and Cardiology. We believe sound analysis will provide a useful yet inexpensive tool for primary care physicians as well as musculoskeletal specialists.

Phase 1: Establish the normal sound patterns emanating from the uninjured knee; we will look for the influence of age, height and weight.

Phase 2: To record and analyze the preoperative sound patterns from the knees with pathology, known by MRI and arthroscopy, then compare them with the normal sounds from Phase 1.

ELIGIBILITY:
Inclusion Criteria:

Phase I

* Healthy Individuals.
* No neurological problems.
* No knee complaints.
* No previous Surgery or Knee injuries.

Phase II Patients undergoing knee arthroscopy who have pre-op MRI. The inclusion will be based on age group, 20 years of age, 40 and 60.

Exclusion Criteria:

* Neurologic Disease
* Previous serious injury (Fracture or dislocation).
* Previous Ligament reconstruction.
* Major non-subtitle problems with their knees. (This would create overwhelming noises).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male or female english-speaking from the ages of 18 thru 70
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-01-20 (Estimated); Primary Completion 2018-02-18 (Estimated); Study Completion 2018-05-18 (Estimated)

PRIMARY OUTCOMES:
Analysis of Joint Sounds in the Diagnosis of Knee Disorders | 1 -2 years
  Phase 1: Analysis will be carried out on the recording from apparently normal knees, sounds are amplification, wave form and filtering. Effects of age, height and weight. Phase 2: analysis of sound will br carried out by a researcher blinded to the MRI and arthroscopic pathology, Then, comparison of the abnormal sounds to the pathology found on the MRI and Arthroscopy to look for correlations.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ludloff D. ie Auskultation der Wirbelsäule, des Kreuzbeins und des Reckens. Münchener medizinische wochenschrift, LIII, 1197, 1906. Walters CF. The Value of Joint Auscultation. In: The Lancet, 1:920-921. 1929. Rangayyan RM, Wu YF. Screening of Knee-Joint Vibroarthrographic Signals Using Statistical Parameters and Radial Basis Functions. In: Medical & Biological Engineering & Computing 46 (3) 2008: pp. 223-232. Chu ML, Gradisar IA, Zavodney LD. Possible Clinical Application of a Noninvasive Monitoring Technique of Cartilage Damage in Pathological Knee Joints. In: Journal of Clinical Engineering 3 (1), 1978: pp. 19-27. McCoy GF, McCrea JD, Beverland DE, Kernohan WG, Mollan RAB. Vibration Arthrography as a Diagnostic Aid in Diseases of the Knee. In: The Journal of Bone and Joint Surgery 69-B (2), 1987: pp. 288-293. Reddy NP, Rothschild BM, Mandal, M, Gupta V, Suryanarayanan S. Noninvasive Acceleration Measurements to Characterize Knee Arthritis and Chondromalacia. In: Annals of Biomedical Engineering, v. 23, pp. 78-84, 1995. Krishnan S, Rangayyan RM, Bell GD, Frank CB, and Ladly KO. Adaptive Filtering, Modeling, and Classification of Knee Joint Vibroarthrographic Signals for Noninvasive Diagnosis of Articular Cartilage Pathology. In: Medical and Biological Engineering and Computing, 35(6):677-684, 1997.